CLINICAL TRIAL: NCT01670630
Title: A Comparison of a Novel Sheathed Speculum to a Standard Speculum for Visualization of the Cervix
Brief Title: A Comparison of a Sheathed to a Standard Speculum for Visualization of the Cervix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: MDI Worldwide LLC (Unknown)
Responsible Party: Principal Investigator, D. Ashley Hill, MD, Associate Director, Department of Obstetrics and Gynecology, Florida Hospital Graduate Medical Education, AdventHealth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CS201202
Record Dates: First submitted 2012-08-07; First posted 2012-08-22 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-02

CONDITIONS: Comparison of a Sheathed Versus Standard Plastic Speculum
Keywords: speculum; vagina; cervix; examination
MeSH Terms: interventions — Surgical Instruments; Condoms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sheathed speculum (Active Comparator): Investigators will perform a vaginal speculum examination with either a sheathed or a standard ("non sheathed" speculum in a randomized comparison to estimate the degree of cervical visualization and subject pain perception.
  Interventions: Procedure: Sheathed speculum examination
- Standard speculum examination (Active Comparator): Investigators will perform a vaginal speculum examination with either a standard or a sheathed speculum in a randomized comparison to estimate the degree of cervical visualization and subject pain perception.
  Interventions: Procedure: Standard speculum examination

INTERVENTIONS:
Procedure: Sheathed speculum examination
  Other Names: speculum; sheath; ClearSpec
  Arms: Sheathed speculum
Procedure: Standard speculum examination
  Arms: Standard speculum examination

SUMMARY:
The purpose of this study is to estimate if a novel sheathed speculum provides improved visualization of the cervix compared to a standard ("non sheathed") speculum, and to estimate if the sheathed speculum causes less discomfort during the examination.

DETAILED DESCRIPTION:
This is a randomized trial where physician investigators will perform clinically indicated vaginal speculum examinations using either a sheathed or a standard plastic speculum, to determine which speculum provides the best visualization of the cervix. As a secondary outcome, study participants will record their pain level on a 10-cm visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing clinically indicated vaginal speculum examination.
* Subject has had at least 1 prior vaginal deliver > 20 weeks gestational age.
* Able to read and speak English.

Exclusion Criteria:

* Active vulvar lesions or conditions (sexually transmitted infections, vestibulodynia, candida, vaginitis, or vulvar dermatologic condition).
* Menopausal or using hormone replacement therapy.
* Genital atrophy.
* Chronic pelvic pain, dyspareunia, or interstitial cystitis.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Degree of cervix visualized. | During vaginal speculum examination.
  To compare the degree of cervical visualization as interpreted by the investigator between the sheathed speculum and the standard plastic disposable speculum.

SECONDARY OUTCOMES:
Comparison of pain during speculum examination. | During speculum examination.
  To compare the subjects' comfort level between the sheathed and standard speculums when undergoing a vaginal speculum examination, using a patient-reported 10-cm visual analog scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: David A Hill, M.D., Principal Investigator — AdventHealth
Locations (1):
- Loch Haven Ob/Gyn Group, Orlando, Florida, United States

REFERENCES:
- [Derived] Hill DA, Cacciatore ML, Lamvu G. Sheathed versus standard speculum for visualization of the cervix. Int J Gynaecol Obstet. 2014 May;125(2):116-20. doi: 10.1016/j.ijgo.2013.10.025. Epub 2014 Feb 1. PMID 24565103